CLINICAL TRIAL: NCT05165511
Title: Executive Function Enhanced Parent-Based Treatment for Children With ADHD and Overweight or Obesity
Brief Title: Families, Responsibility, Education, Support, and Health for Executive Function
Acronym: FRESH-EF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Rady Children's Hospital, San Diego (Other)
Responsible Party: Principal Investigator, Dawn Eichen, Assistant Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 210123
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Overweight and Obesity; Attention-Deficit Hyperactivity Disorder
Keywords: weight loss; executive function; parent-based treatment
MeSH Terms: conditions — Overweight; Obesity; Attention Deficit Disorder with Hyperactivity; Weight Loss

STUDY DESIGN:
Intervention Model Description: This is an open-label one-arm pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Executive Function-Enhanced Parent-Based Behavioral Treatment (PBT-EF) (Experimental): PBT-EF will integrate executive function training with family-based behavioral treatment (FBT) for obesity, the gold-standard behavioral treatment for childhood obesity. PBT-EF will include self-monitoring, calorie reduction, and dietary and physical activity recommendations in addition to planning, organization, and problem-solving skills.
  Interventions: Behavioral: PBT-EF

INTERVENTIONS:
Behavioral: PBT-EF — PBT-EF will be delivered to parents only. Parents will be taught general behavioral weight loss skills to apply to their child and themselves including decreasing caloric intake and increasing physical activity, self-monitoring, and goal setting. Additionally, parents will learn compensatory strategies surrounding organization, habit learning, planning, and problem-solving to generalize FBT skills to real-world behaviors (e.g., self-monitoring of food intake). Each session will include interactive exercises to help train an aspect of EF. Skills taught will be presented to be practiced with real-world applications.

SUMMARY:
The pilot study will be a one group open-label treatment program and will be used to refine a parent-based behavioral treatment enhanced with executive-function training (PBT-EF) for children with comorbid overweight or obesity and Attention-Deficit Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
The currently recommended treatment for children with overweight or obesity (OW/OB), family-based behavioral treatment (FBT), results in sustained weight loss for only 1/3 of children. Attention-Deficit Hyperactivity Disorder (ADHD) is one of the most common neurobehavioral disorders in children and is characterized by difficulties in Executive Function (EF). Substantial research suggests higher rates of OW/OB in children with ADHD; thus, children with OW/OB and ADHD are likely to have greater difficulties with EF and achieving success in FBT. The proposed study aims to develop a parent-based behavioral treatment enhanced with EF training (PBT-EF) to improve treatment outcomes for children with comorbid OW/OB and ADHD. The treatment will be administered to parents in 18 group sessions over 5 months. Parents and children will be assessed at baseline, post-treatment, and 3-month follow-up. Assessments will include body mass index (BMI), assessments of executive function, and behavioral questionnaires. This study could provide a novel model to treat OW/OB in children with ADHD, and could inform clinical decision making regarding obesity treatment.

ELIGIBILITY:
Inclusion Criteria:

* Child with overweight or obesity (85-99.9% BMI for age),
* Child age 8-12,
* Child with a diagnosis of ADHD,
* A parent willing to participate who can read and understand English at a minimum of a fifth-grade level, able to attend treatment sessions remotely via Zoom on video.

Exclusion Criteria:

* Current enrollment in an organized weight control program (parent and child)
* Medication specifically prescribed for weight loss (child)
* Medical or psychiatric condition that may interfere with treatment participation or that may require physician monitoring of diet and/or exercise (e.g., acute suicidality; psychosis; substance use disorder) (parent and child)
* Change in psychotropic medication or other medication that may impact weight or ADHD symptoms during the previous 3 months (child)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility as measured by number of treatment sessions attended | Over the course of 5 months of treatment
  Attendance at Treatment Sessions
Acceptability | At 5 months
  Ratings of usefulness of treatment

OTHER OUTCOMES:
Child body mass index (BMI) | Change from baseline at an average of 5 months and 8 months
  As measured by height and weight (kg/m^2)
Child executive function | Change from baseline at an average of 5 months and 8 months
  Change in executive function measured by Behavior Rating in Executive Functioning - 2 (BRIEF-2). The Global Executive Composite score reflects a standardized t-score with higher scores reflecting greater difficulties in executive function.
Parent executive function | Change from baseline at an average of 5 months and 8 months
  Change in executive function measured by Behavior Rating in Executive Functioning - Adult (BRIEF-A). The Global Executive Composite score reflects a standardized t-score with higher scores reflecting greater difficulties in executive function.
Child behavioral symptoms - Child Behavior Checklist (CBCL) | Change from baseline at an average of 5 months and 8 months
  Change in child behavioral symptoms rated by parents as measured by CBCL. The CBCL is a widely used parent-report questionnaire designed to assess behavioral problems and social competencies of children ages 4-18. It yields standardized T scores and age adjusted scores on internalizing, externalizing, and total behavior difficulties. Higher scores reflect greater behavioral difficulties.
Child behavioral symptoms - Vanderbilt ADHD [Attention Deficit Hyperactivity Disorder] Parent Rating Scale | Change from baseline at an average of 5 months and 8 months
  Change in child behavioral symptoms rated by parents as measured by Vanderbilt ADHD Parent Rating Scale. This scale is a parent-report questionnaire. The parent rates the frequency of 47 behaviors that may indicate behavioral issues. There are also 8 performance questions. Change in total symptoms of the 18 ADHD criteria will be reported. Higher scores reflect greater ADHD symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn M Eichen, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Center for Healthy Eating and Activity Research (CHEAR), San Diego, California, United States